CLINICAL TRIAL: NCT01981655
Title: A Phase 2, Randomised, Single-Blind, Placebo-controlled Study of Half Molar Sodium Lactate Solution in the Treatment of Subjects With Acute Heart Failure
Brief Title: 0.5M Na Lactate Solution in Acute Heart Failure (AHF)
Acronym: SOLACE1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nepean Blue Mountains Local Health District (Other)
Collaborators: Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Principal Investigator, Marek Nalos, Staff Specialist, Intensive Care Medicine, Nepean Blue Mountains Local Health District
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOLACE1
Record Dates: First submitted 2013-08-13; First posted 2013-11-11 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Acute Heart Failure
Keywords: Sodium Lactate; Acute; Heart; Failure; Perfusion
MeSH Terms: interventions — Sodium Lactate; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5M Sodium lactate (Experimental): A bolus of 0.5M Sodium lactate of 3 ml per kg body weight (BW) is administered in 15 minutes, followed by a continuous infusion with 1 ml per kg per hour for 24 hours, i.e. in total 27 ml per kg over 24 hours
  Interventions: Drug: 0.5M Sodium lactate
- Hartmann's solution (Active Comparator): Hartmann's solution of 3 ml per kg BW is administered in 15 minutes. There is NO continuous infusion infused thereafter; i.e. in total 3 ml per kg over 24 hours
  Interventions: Drug: Hartmann's solution

INTERVENTIONS:
Drug: 0.5M Sodium lactate — A bolus of 0.5M Sodium lactate of 3 ml per kg BW is administered in 15 minutes, followed by a continuous infusion with 1 ml per kg per hour for 24 hours, i.e. in total 27 ml per kg over 24 hours
  Other Names: Totilac
  Arms: 0.5M Sodium lactate
Drug: Hartmann's solution — Hartmann's solution of 3 ml per kg BW is administered in 15 minutes, No infusion thereafter i.e. in total 3 ml per kg over 24 hours
  Other Names: Compound Sodium Lactate
  Arms: Hartmann's solution

SUMMARY:
The objective of this trial to see whether:

-Cardiac performance (cardiac index and secondary outcomes)can be improved in patients with acute heart failure (AHF) and symptoms and consequences of fluid overload (pulmonary and interstitial edema) and poor peripheral perfusion can be reduced by:

1. Providing lactate as a substrate(Improve cardiac index)
2. Simultaneously restoring optimal preload

Optimal standard treatment will be achieved in both arms with the use of current best treatment protocol for AHF as per independent treating physician.

4. To assess effects of 0.5M Na lactate (Totilac) on plasma and urine biological parameters (sodium, potassium, chloride, pH, bicarb, base excess, albumin)

5. To assess effects of 0.5M Na lactate on morbidity and mortality.

DETAILED DESCRIPTION:
* Acute heart failure is a critical illness for which current treatments are suboptimal.
* The various symptoms are related to inadequate cardiac output and usually include left ventricular overload with pulmonary oedema, interstitial fluid accumulation and tissue oedema (as indicated by frequent hyponatremia and hypoalbuminemia) and insufficient peripheral perfusion frequently manifesting as cold extremities and low urine output.
* The current treatment of this syndrome is based on diuretics, vasodilators and/or inotropes, but fluid administration is also required to optimise the intravascular volume state and to reverse shock if present. Therefore management of body fluid balance remains a challenge since treatment aims to simultaneously maintain or improve intravascular volume and decrease body fluid excess and oedema.
* The purpose of the present study is to assess in a prospective randomised trial the efficacy and safety of a newly designed crystalloid solution, 0.5 M sodium lactate, with properties potentially able to improve multiple pathophysiological aspects of AHF, as compared to the use of standard crystalloid solution Compound Sodium Lactate (mildly hypoosmolar ~ 274 mOsm/L and isotonic).

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 18 years
* Heart failure criteria:

Left heart failure: as evidenced by 2 out of 3:

* Left ventricular ejection fraction (LVEF) ≤ 40% and cardiac index ≤ 2.5 L/min/m2
* Acute pulmonary oedema of cardiac origin or mechanical ventilation (including CPAP/BIPAP) for respiratory failure of predominantly cardiac origin
* Need for inotropes/vasopressors for cardiac pump failure OR

Right heart failure: as evidenced by 1 out of 2:

* Bilateral leg oedema above ankles
* RV failure (low tricuspid annular plane systolic excursion (TAPSE), dilated floppy RV)
* Poor peripheral perfusion as evidenced by 2 out of 3:

Cold mottled skin Low urine output Acutely clouded sensorium/poor mentation

* Consent obtained from patient or patient's next of kin.

Exclusion Criteria:

* Hypernatremia: [Na] >145 mmol/L
* Diagnosed hypertrophic obstructive cardiomyopathy
* Uncorrected severe valvular heart disease
* Documented third degree heart block, sustained ventricular tachycardia
* Documented cardiac tamponade
* Septic shock
* Acute respiratory distress syndrome (ARDS)
* Moribund patients likely to die before 24h
* Patients with major diseases of limited prognosis such as end stage cancer,end-stage liver failure, end stage dialysis dependent renal failure
* Patients with absolute indication for acute hemodialysis/hemofiltration (pH, K, urea > 35 mmol/L, severe fluid overload in the presence of oliguria < 200 mL/6h.
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | Baseline till 24 hours from first loading of study drug
  Improvement in cardiac output measured by transthoracic echocardiography at 24 hours from initiation of study drug infusion

SECONDARY OUTCOMES:
mortality | up to 3 month
  range of efficacy and safety parameters
acid base and electrolytes, fluid balance | 48 hours
  the effect on on pH, base excess, bicarbonate, sodium, potassium, phosphate, chloride and lactate will be assessed during the study period
organ function | 48 hours
  effect on respiratory function assessed by time on ventilatory support and renal function measured by creatinine level over 48 hours will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Marek Nalos, MD, Principal Investigator — Dept. of Intensive Care, Nepean Hosp., U Sydney, Penrith, NSW, Australia
Locations (1):
- Dept. of Intensive Care, Nepean Hosp., U Sydney, Penrith, New South Wales, Australia

REFERENCES:
- [Derived] Nalos M, Leverve X, Huang S, Weisbrodt L, Parkin R, Seppelt I, Ting I, Mclean A. Half-molar sodium lactate infusion improves cardiac performance in acute heart failure: a pilot randomised controlled clinical trial. Crit Care. 2014 Mar 25;18(2):R48. doi: 10.1186/cc13793. PMID 24666826